CLINICAL TRIAL: NCT00656123
Title: A Safety and Feasibility Study of an Allogeneic Colon Cancer Cell Vaccine Administered With a GM-CSF Producing Bystander Cell Line in Patients With Metastatic Colorectal Cancer
Brief Title: Study of Colon GVAX and Cyclophosphamide in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0745; NA_00009345
Record Dates: First submitted 2008-04-09; First posted 2008-04-10 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CY and colon GVAX (Experimental)
  Interventions: Biological: Colon GVAX; Drug: cyclophosphamide

INTERVENTIONS:
Biological: Colon GVAX — Dose escalation: 1.4x10^8 to 7x10^8 cells administered in up to 15 intradermal injections on Day 2 of Cycles 1-4
  Other Names: Allogeneic Colon Cancer Cell Vaccine Administered with a Granulocyte-Macrophage Colony Stimulating Factor-Producing Bystander Cell Line
Drug: cyclophosphamide — 200 mg/m^2 administered IV on Day 1 of Cycles 1-4

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of vaccination with two irradiated allogeneic colorectal carcinoma cells administered with a GM-CSF producing bystander cell line in sequence with an immunomodulatory dose of Cyclophosphamide

ELIGIBILITY:
Inclusion Criteria:

* Documented metastatic colorectal cancer
* ECOG Performance Status of 0 to 1
* Adequate organ function as defined by study-specified laboratory tests
* Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
* Signed informed consent form
* Life expectance > 12 weeks

Exclusion Criteria:

* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune, or other medical conditions
* Systemically active steroid use
* Another investigational product within 28 days prior to receiving study drug
* Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug
* Chemotherapy, radiation, or biological cancer therapy within 28 days prior to receiving study drug
* No known history or evidence of CNS metastases < 2 years.
* Pregnant or lactating
* Unwilling or unable to comply with study procedures

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients Experiencing a Grade 3 or Above Treatment-related Toxicity | 3.5 years
  When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v3) will be counted only once for a given subject.

SECONDARY OUTCOMES:
Percent Fold change in amount of interferon gamma-producing Ep-CAM-specific CD8 T cells after vaccination | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng L, Edil BH, Soares KC, El-Shami K, Uram JN, Judkins C, Zhang Z, Onners B, Laheru D, Pardoll D, Jaffee EM, Schulick RD. A safety and feasibility study of an allogeneic colon cancer cell vaccine administered with a granulocyte-macrophage colony stimulating factor-producing bystander cell line in patients with metastatic colorectal cancer. Ann Surg Oncol. 2014 Nov;21(12):3931-7. doi: 10.1245/s10434-014-3844-x. Epub 2014 Jun 19. PMID 24943235